CLINICAL TRIAL: NCT07119073
Title: An Open-label, Randomized, Single-dose, Two-period, Two Treatment (Fed vs Fasted), Two Sequence, Crossover Study in Healthy Adult Subjects to Assess the Effect of Food on the Bioavailability of CTx-1301 (Dexmethylphenidate)
Brief Title: In-clinic Crossover Study in Subjects With Two Treatments (Fed vs Fasted)
Acronym: Fed-Fast
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cingulate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CTx-1301-013
Record Dates: First submitted 2025-04-25; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers in Fed and Fasted State
Keywords: Healthy Normal Volunteers; Fed Study; Pharmacokinetics; Dexmethylphenidate; Bioavailability; d-MPH; dMPH
MeSH Terms: conditions — Fasting | interventions — Dexmethylphenidate Hydrochloride

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to one of two sequences: Sequence 1) Fasted:Fed or Sequence 2) Fed:Fasted
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CTx-1301 Fasted (Active Comparator): Subjects will receive CTx-1301 in a fasted state
  Interventions: Drug: Dexmethylphenidate
- CTx-1301 Fed (Active Comparator): Subjects will receive CTx-1301 in a fed state (high fat test meal)
  Interventions: Drug: Dexmethylphenidate

INTERVENTIONS:
Drug: Dexmethylphenidate — Subjects will be randomized to one of two sequences. Subjects will be dosed with 50 mg dose of Cox-1301 during each sequence. Subjects will serve as their own control.

SUMMARY:
The primary purpose of this study is to assess the effect of food on the rate and extent of absorption and the overall bioavailability of a single dose of CTx-1301 50 mg trimodal tablets in healthy adult volunteers.

DETAILED DESCRIPTION:
Fasted Arm: Following an overnight fast of at least 10.5 hours prior to dosing, subjectsshould be administered CTx-1301 (50 mg) with approximately240 mL (8 fluidounces) of water. No food should be allowed for at least 4 hours post-dose.Water can be allowed as desired except for at least one hour before and at least one hour after drug administration. Subjects should receive standardized meals as defined in the study schedule for the fasted treatment arm.

Fed Arm: Following an overnight fast of at least 10.5 hours prior to dosing, subjects should begin consuming the test meal 30 minutes prior to administration ofCTx-1301. CTx-1301 (50 mg) should be administered 30 minutes after thestart of the meal. CTx-1301 (50 mg) should be administered with approximately240 mL (8 fluid ounces) of water. No food should be allowed for at least 4 hours post-dose. Water can be allowed as desired except for at leastone hour before and at least one hour after drug administration. Subjects will receive the high-fat meal as described below for the fed treatment arm and standardized meals for all other meals.

A high-fat (approximately 50 percent of total caloric content of the meal) and high-calorie (800 to 1000 calories) meal is used as the test meal for food-effect bioavailability (BA) and fed bioequivalence (BE) studies. This test meal allows 150, 250, and 500-600 calories from protein, carbohydrate, and fat, respectively. The test meal must be entirely consumed within 30 minutes prior to administration of CTx-1301; the test meal consists of two eggs fried in butter, two strips of bacon, two slices of toast with butter, four ounces of hash brown potatoes and eight ounces of whole milk.

ELIGIBILITY:
Inclusion Criteria:

1. Gender

   a. Male or Female
2. Age

   1. Aged between 18 and 50 years inclusive. Weight and BMI

   <!-- -->

   1. Body weight ≥ 50 kg
   2. BMI ≥ 18 and ≤ 30

4. Compliance

1. Understands and is willing, able, and likely to comply with all study procedures and restrictions.
2. Able to fully consume the required fed meal within 30 minutes without substitutions.
3. If sexually active, male subjects must use an acceptable method of contraception, which includes the double-barrier method (condom and spermicide) or agree to remain abstinent from heterosexual intercourse from Qualification day, during the study, and for 90 days following the last administration of study drug.
4. If sexually active, female subjects of child-bearing potential must use an acceptable method of contraception, which includes, hormonal contraceptives, intrauterine device (IUD) with or without hormones, or double-barrier method (e.g. condom and spermicide), or remain abstinent from heterosexual intercourse for 30 days prior to screening during the study and for 30 days following the last administration of study drug.
5. Male subjects must agree not to donate sperm during the study and for 90 days following the last administration of study drug.
6. Female subjects must agree not to donate eggs during the study and for 30 days following the last administration of study drug.

   5. Consent

a. Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent (signed and dated) obtained before any study-related activities are performed.

6. General Health

1. Good general health (in the opinion of an investigator) with no clinically significant or relevant abnormalities on medical history, laboratory results, or physical examination which could affect the safety of the subject or integrity of study data.
2. No signs of illness (fever or vomiting) within 24-hours of admission on Qualification day and check-in at Day -1
3. Subject has sufficient venous access at the time of screening to allow cannulation and/or venipuncture to obtain the required volume of blood for this study.

   7. Smoking/Caffeine/Alcohol

<!-- -->

1. Subject must be a non-smoker (i.e., does not use any form of nicotine products) as defined by exclusion #4 in this protocol.
2. Subject must be able to refrain from caffeine or xanthine-containing beverages or foods (e.g., tea, coffee, chocolate, cola) for 24 hours prior to admission on Qualification day, check-in at Day -1 and for the duration of the stay at the study center until EOS.
3. Subject must be able to refrain from using alcohol 48 hrs. prior to admission on Qualification day, check-in at Day -1 and for the duration of the stay at the study center until EOS.

   8. Medications

a. Subject must be willing and able to take stimulant medications during participation in this trial.

9. Qualification

a. Subject satisfactorily completes the Qualification day, is able to safely tolerate 30 mg Focalin™ XR, and general behavior suggests that the subject could successfully complete the study in the opinion of an investigator.

Exclusion Criteria:

1. Medical History

   1. Current and/or recurrent disease or illness that, in the opinion of an investigator, could affect the study conduct, study outcome, subject safety, or pharmacokinetic (PK) assessments (e.g., hepatic disorders, renal insufficiency, non-self-limiting gastrointestinal disorders, weight loss surgeries).
   2. Any clinically significant history including but not limited to arterial hypertension, pulmonary arterial hypertension, myocardial infarction, peripheral vascular disease, stroke, or evidence of other cardiovascular disease or disorder, including but not limited to ECG abnormalities such as:

      • QT interval measurement corrected for heart rate according to the Fridericia rule (QTcF) >450 msec for males or >470 msec for female subjects during controlled rest at screening, qualification, and Day -1,

      • Family history of long QT syndrome,

      • Family history of congenital QT prolongation,

      • PR (PQ) interval shortening <120 msec (PR <120 msec but >110 msec is acceptable if there is no evidence of ventricular pre-excitation),

      • PR (PQ) interval prolongation (>220 msec), intermittent second-degree (Wenckebach block while asleep or in deep rest is not exclusionary), or third-degree atrioventricular block,

      • Persistent or intermittent complete bundle branch block (BBB) or intraventricular conduction delay (IVCD) with QRS >110 msec.
   3. Current and/or previous history of any other serious, severe or unstable psychiatric illness which in the opinion of the investigator, may require treatment (e.g. anxiety, psychosis, mood disorder, motor tics or suicidality) or make the subject unlikely to fully complete the study, and/or any condition that presents undue risk from the study medication or procedures.
   4. Subject has had suicidal thoughts within the last 6 months as supported by the Columbia Suicide Severity Rating Scale (C-SSRS).
   5. Positive test results for Human Immunodeficiency Virus (HIV)-1/HIV-2 antibodies, Hepatitis B surface antigen (HBsAg) or Hepatitis C virus antibody (HCVAb).
   6. A family history of sudden cardiac or unexplained death.
   7. Any condition or abnormal laboratory finding that could result in harm to the subject, affect the outcome of the study or suggest unstable medical illness.
   8. Any clinically significant psychiatric disorder or finding which the Investigator considers the subject disqualified from the study.
   9. Subject plans to undergo elective procedures/surgery at any time during the study.
   10. Subject has had surgery within the past 90 days.
   11. Subject of child-bearing potential is pregnant or planning to become pregnant during the duration of the study or within 30 days of the end of the study.
   12. Subject is breast-feeding during the study or within 30 days following the study.
2. Medications a. Subject has taken any medication that, in the opinion of an Investigator, has been shown to alter the PK of d-MPH.

   b. Use of any prescription medication within 14 days prior to Qualification and Day -1 and/or use of any OTC medications (such as antacids, vitamins, minerals, dietary/herbal preparations, and nutritional supplements) within 7 days prior to Qualification and Day -1, unless jointly approved by an Investigator and Sponsor. Subjects may not use these medications for the full duration of the stay at the study center until EOS.

   i. Subjects are permitted to take hormonal contraceptives and hormone replacement therapy at acceptable levels if stable at least 30 days prior to Qualification, through the duration of the study, and for 30 days after the study ends.

   ii. Acetaminophen (up to 2 grams per day) may be used during the study under the direction of the Investigator.

   iii. COVID vaccine is allowed if taken at least 45 days prior to Qualification Protocol CTx-1301-013 Version 1.0 Page 25 of 49 CONFIDENTIAL iv. On a case-by-case basis, an Investigator is permitted to allow the use of certain concomitant medications, for example, to treat an AE, as long as an Investigator determines that the medication will not affect the subject's safety or study integrity (e.g., topical medications).
3. Alcohol/Substance Abuse

   a. Lifetime history of alcohol or other substance abuse. b. Subject has positive urine alcohol test or urine screen for drugs of abuse at screening, qualification or check-in. (Screening visit urine MPH screen results are not required prior to Qualification day but are necessary prior to randomization on Day -1. Day-1 urine MPH screen results are not required prior to dosing in each Period).
4. Smoking

   a. Subject is a current smoker or has recently discontinued smoking (i.e., regular use of any nicotinecontaining products within 3 months of screening). Occasional, social use, or routine environmental exposure to nicotine is acceptable.
5. Allergy/Intolerance

   a. Subject has a history of allergy to d-MPH, to any component of the dosage form, or any other allergy, which, in the opinion of an Investigator, contraindicates their participation.
6. Clinical Studies

   a. Receipt of an investigational drug within the 30 days before screening day. b. Previous participation in a CTx-1301 study.
7. Personnel

   a. An employee of the sponsor, study site, or members of their immediate family.
8. Blood

   1. Subject has donated blood within 56 days prior to screening, plasma within 7 days prior to screening, or experienced significant blood loss (excess of 500 mL) within 3 months prior to screening and for the duration of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2024-10-31 (Actual); Primary Completion 2024-12-21 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter (Cmax) | Hour 0 to hour 28
  Maximum Concentration
Pharmacokinetic parameter (AUC0-inf) | Hour 0 to hour 28
  Area Under the Curve from time 0 to infinity
Pharmacokinetic parameter (AUC0-last) | Hour 0 to hour 28
  Area Under the Curve from time 0 to 28 hrs

SECONDARY OUTCOMES:
Pharmacokinetic parameter K | Hour 0 to hour 28
  Terminal Elimination Constant
Pharmacokinetic parameter T 1/2 | Hour 0 to hour 28
  Half Life
Pharmacokinetic parameter T max | Hour 0 to hour 28
  Time of Maximum Concentration
Pharmacokinetic parameter T lag | Hour 0 to hour 28
  Lag time
Pharmacokinetic parameter Cl/F | Hour 0 to hour 28
  Apparent Clearance
Pharmacokinetic parameter Vd/F | Hour 0 to hour 28
  Apparent Volume of Distribution
Partial AUC | 0-3 hrs
  Area Under the Curve
Partial AUC | 3-6 hrs
  Area Under the Curve
Partial AUC | 3-7 hrs
  Area Under the Curve
Partial AUC | 6-9 hrs
  Area Under the Curve
Partial AUC | 7-12 hrs
  Area Under the Curve
Partial AUC | 9-12 hrs
  Area Under the Curve
Partial AUC | 12-16 hrs
  Area Under the Curve
Safety - ECG | Day -1 to Day 4
  Evaluation of changes in ECG measurements; heart rate, PR interval, RR interval, QT interval, QTc with Bazett correction, QTc with Fredericia correction intervals, and QRS duration.
Safety - Vital Signs | Day -1 to Day 4
  Evaluation of changes in Vital Sign measurements to include blood pressure (mmhg).
Safety - Vital Signs | Day -1 to Day 4
  Evaluation of changes in Vital Sign measurements to include weight (kg).
Safety - Vital Signs | Day -1 to Day 4
  Evaluation of changes in Vital Sign measurements to include heart rate (bpm).
Safety - Vital Signs | Day -1 to Day 4
  Evaluation of changes in Vital Sign measurements to include height (cm).
Safety - Vital Signs | Day -1 to Day 4
  Evaluation of Vital Sign measurements to include weight and height combined to report BMI in kg/m^2.
Safety - Safety Labs | Day -1 to Day 4
  Evaluation of changes in Safety Lab measurements to include hematology, biochemistry, thyroid, serology, urinalysis, and drugs of abuse.
Safety - Physical Exam | Day -1 to Day 4
  Evaluation of changes in the Physical Exam to include general appearance, skin, head, eyes, ears, nose, throat, neck, spine, psychiatric, respiratory, cardiovascular, gastrointestinal, musculoskeletal, central nervous system, lymphatic, endocrine.
Safety - C-SSRS | Day -1 to Day 4
  C-SSRS is a tool designed to access and track suicidal adverse events (suicidal behavior and suicidal ideation).
Safety - Treatment Emergent Adverse Events (TEAEs) | Day -1 to Day 4
  Evaluation of Treatment Emergent Adverse Events (TEAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Matt Brams, MD, Study Director — Cingulate Therapeutics
Locations (1):
- Dr. Vince Clinical Research, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No